CLINICAL TRIAL: NCT04830579
Title: Randomized Crossover Two Period Single Dose Bioequivalence Study of Two Formulations Etoricoxib Tablets 120 mg (Pharmtechnology LLC, Republic of Belarus) and Arcoxia® Tablets 120 mg (Merck Sharp & Dohme B.V., Netherlands) in Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Two Formulations of Etoricoxib Tablets 120 mg in Healthy Volunteers Under Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: ClinPharmInvest, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ETRXB-2020-CPI-FRMT
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Bioequivalence
Keywords: Etoricoxib; Bioequivalence; Arcoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence TR (Other): 17 subjects assigned to the sequence TR will receive a single 120 mg dose of the test product Etoricoxib (1 x 120 mg tablet), marked as T in the sequence, in Period 1 and a single 120 mg dose of the reference product Arcoxia® (1 x 120 mg tablet), marked as R in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Etoricoxib film-coated tablet 120 mg; Drug: Arcoxia® film-coated tablet 120 mg
- Sequence RT (Other): 17 subjects assigned to the sequence RT will receive a single 120 mg dose of the reference product Arcoxia® (1 x 120 mg tablet), marked as R in the sequence, in Period 1 and a single 120 mg dose of the test product Etoricoxib (1 x 120 mg tablet), marked as T in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Etoricoxib film-coated tablet 120 mg; Drug: Arcoxia® film-coated tablet 120 mg

INTERVENTIONS:
Drug: Etoricoxib film-coated tablet 120 mg — Etoricoxib is manufactured by Pharmtechnology LLC, Republic of Belarus. Each tablet contains 120 mg of etoricoxib.
  Other Names: The test product
Drug: Arcoxia® film-coated tablet 120 mg — Arcoxia® is manufactured by Frosst Iberica SA, Spain. Each tablet contains 120 mg of etoricoxib.
  Other Names: The reference product

SUMMARY:
This is an open-labeled, randomized, two period, single-center, crossover, comparative study, where each participant will be randomly assigned to the reference (Arcoxia®, 120 mg film-coated tablets) or the test (Etoricoxib, 120 mg film-coated tablets) formulation in each period of study (sequences Test-Reference (TR) or Reference-Test (RT)), in order to evaluate if both formulations are bioequivalent.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy caucasian men or women aged between 18 to 45 years 2. Verified diagnosis "healthy" according to the anamnesis data and the results of standard clinical, laboratory and instrumental examination methods, physical examination and anamnestic examination 3. The results of an X-ray or fluorographic examination of the chest organs within the normal range (the results of an examination carried out within 12 months before the start of the study may be provided) 4. Body mass index 18.5-30 kg/m² 5. For female subject:

* the results of the examination of the mammary glands (palpation or mammography) within the normal range according to the data obtained within 12 months before the start of the study,
* Non-breastfeeding women,
* Non-pregnant women (negative pregnancy test),
* If subject is a female and is of childbearing potential, she should be practicing an acceptable method of birth control for the duration of the study (the entire time from at least 14 days before taking the drug in the first period and within 14 days after taking the drug in the second period): sexual continence, or condom + spermicide, or diaphragm + spermicide. Intrauterine contraception is also a reliable method of contraception, installed at least 4 weeks before taking the study drugs in the first period,
* women who are not using acceptable methods of contraception if they are considered incapable of childbearing can participate in the study: women who have undergone a hysterectomy or tubal ligation, women with a clinical diagnosis of infertility, and women who are in menopause (at least a year without menstruation in the absence of alternative medical conditions),
* in case of using contraceptives (injectable and oral hormonal contraceptives, subcutaneous hormonal implants or intrauterine hormonal therapeutic systems), the latter should be canceled at least 60 days before taking the drug in the first period; 6. Consent to use a double barrier method of contraception (condom + spermicide) or sexual continence, as well as consent not to take part in sperm donation from the moment of taking the drug in the first period, during the entire study and within 14 days after taking the drug in the second period research 7. Subjects are able to understand the requirements of the study, to sign a written informed consent, and also to accept all the restrictions imposed during the course of the study, and to agree to return for the required investigations

  1. Burdened allergic history, hypersensitivity to etoricoxib or excipients that are part of any of the investigational drugs, or intolerance to these components.
  2. Complete or incomplete combination of bronchial asthma, acute rhinitis, recurrent polyposis of the nose and paranasal sinuses and intolerance to acetylsalicylic acid or intolerance to other NSAIDs (including a history).
  3. Increased risk of complications from the gastrointestinal tract due to the use of NSAIDs, peptic ulcer and duodenal ulcer in the acute stage or active gastrointestinal bleeding (including a history).
  4. Hereditary intolerance to lactose or galactose (for example, congenital lactase deficiency or glucose-galactose malabsorption).
  5. Clinically significant pathologies of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys and blood.
  6. Other diseases that, in the opinion of the researcher, may affect the absorption, distribution, metabolism or excretion of both drugs, or increase the risk of negative consequences for the volunteer.
  7. The presence of mental disorders, including a history.
  8. Surgical interventions on the gastrointestinal tract, with the exception of appendectomy.
  9. Acute infectious diseases that ended less than 4 weeks before taking the drug in the first period.
  10. Dehydration due to diarrhea, vomiting or other reason within the last 24 hours before taking the drug in the first period of the study, if vomiting or diarrhea wasn't a manifestation of an infectious disease.
  11. Clinically significant abnormalities on the ECG, the level of systolic blood pressure (SBP) measured in the sitting position at the time of screening <100 mm Hg or ≥ 130 mm Hg and / or diastolic blood pressure (DBP) <60 mm Hg or ≥ 85 mm Hg.
  12. Heart rate less than 60 beats/min or more than 90 beats/min at the time of screening, respiratory rate less than 12 or more than 18 per minute at the time of screening, body temperature below 36.0 ° C or above 37.0 ° C at the time of screening.
  13. Use of any prescription and OTC drugs:

      * including herbs and food additives, vitamins that can have a significant effect on the PK of etoricoxib or data on the effect of which on the pharmacokinetics of etoricoxib are unknown, as well as question the characterization of the volunteer as healthy, less than 14 days before taking the drug in the first period;
      * including the use of drugs that are inducers or inhibitors of isoenzymes CYP3A4 (HIV protease inhibitors, antifungal drugs of the azole group, clarithromycin, erythromycin, phenytoin, carbamazepine, phenobarbital, St. John's wort preparations, etc.), less than 30 days before taking the drug in the first period;
      * the use of injectable and oral hormonal contraceptives, subcutaneous hormonal implants or intrauterine hormonal therapeutic systems for 60 days before taking the drug in the first period.
  14. Donation of plasma or blood (450 ml or more) less than 2 months (60 days) before taking the drug in the first period.
  15. Consumption of caffeine and xanthine-containing drinks and products (tea, coffee, chocolate, cola, etc.), products containing poppy seeds, less than 48 hours before taking the drug in the first period.
  16. Consumption of alcohol and alcohol-containing foods and beverages less than 48 hours before taking the drug in the first period.
  17. Use of citrus fruits (including grapefruit and grapefruit juice) and cranberries (including juices, fruit drinks, etc.) less than 7 days before taking the drug in the first period.
  18. Intake of more than 10 units alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml dry wine or 50 ml of spirits) or history of alcoholism, drug addiction, drug abuse.
  19. Intense physical activity less than 24 hours before taking the drug in the first period.
  20. Smoking more than 10 cigarettes per day, including less than 24 hours before taking the drug in each period and during each study period.
  21. Participation in other clinical trials of drugs less than 3 months before taking the drug in the first period.
  22. Test positive for syphilis, hepatitis B, hepatitis C or HIV at the time of screening.
  23. Positive pregnancy test at screening.
  24. Breastfeeding.
  25. Positive test for alcohol in exhaled air at screening.
  26. Positive urinalysis for the content of narcotic and potent substances during screening (opiates, morphine, barbiturates, benzodiazepines, cannabinoids/marijuana).
  27. The value of standard laboratory and instrumental parameters that go beyond the reference values.
  28. Lack of intention of volunteers to comply with the Protocol requirements throughout the course of the study and/or lack, in the opinion of the Investigator, of the volunteers' ability to understand and evaluate the information on this study as part of the informed consent form signing process, in particular regarding the expected risks and possible discomfort.
  29. Tattooing and piercing within 30 days prior to first drug administration.
  30. Difficulty swallowing tablets.
  31. Difficulty with taking blood (for example, difficult access to the veins).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-04-10 (Estimated); Primary Completion 2021-04-28 (Estimated); Study Completion 2021-04-28 (Estimated)

PRIMARY OUTCOMES:
Cmax of etoricoxib in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00, 96.00 hours after each drug administration.
  Maximum observed concentration in plasma.
AUC0-t of etoricoxib in plasma after administration of the test and the reference. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00, 96.00 hours after each drug administration.
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration (TLQC) using the linear trapezoidal method

SECONDARY OUTCOMES:
Tmax of etoricoxib in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00, 96.00 hours after each drug administration.
  Time of maximum observed concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value.
TLQC of etoricoxib in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00, 96.00 hours after each drug administration.
  Time of last observed quantifiable concentration.
AUC0-INF of etoricoxib in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00, 96.00 hours after each drug administration.
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-t + ĈLQC (the predicted concentration at time TLQC) / λZ (apparent elimination rate constant).
Residual area of etoricoxib in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00, 96.00 hours after each drug administration.
  Extrapolated area (i.e. percentage of AUC0-INF due to extrapolation from TLQC to infinity).
Time point where the log-linear elimination phase begins (TLIN) of etoricoxib in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00, 96.00 hours after each drug administration.
  Time point where the log-linear elimination phase begins.
λZ of etoricoxib in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00, 96.00 hours after each drug administration.
  Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus time curve.
Terminal elimination half-life (Thalf) of etoricoxib in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00, 96.00 hours after each drug administration.
  Terminal elimination half-life, calculated as ln(2)/λZ.
Number of treatment-emergent adverse events for the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00, 96.00 hours after each drug administration.
  The safety population will include all subjects who received at least one dose of the test or the reference product. Any significant changes will be recorded as treatment-emergent adverse events only if they are judged clinically significant by the qualified investigator or delegate.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Khokhlov, Principal Investigator — ClinPharmInvest, LLC
Locations (1):
- Private healthcare institution "Clinical Hospital "RZD-Medicine" of the city of Yaroslavl", Yaroslavl, Russia